CLINICAL TRIAL: NCT07059234
Title: The Motor Activity - Subjective Energy (MASE) Project: Neurobiological and Digital Phenotyping Towards Digital Mental Health Interventions in Depression
Brief Title: The Motor Activity - Subjective Energy (MASE) Project
Acronym: MASE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: University of Salzburg (Other); University of Wuerzburg (Other); University of Mannheim (Other); University of Ostrava (Other); University of Deusto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-00691
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Ambulatory Assessment, Within-Person-Encouragement-Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A, 50% (Experimental): The investigators will compare the physical activity just-in-Time Adaptive Interventions (JITAI) to an active control working memory task within participants. There will be 4 triggers in total. Ratio intervention / active control = 2:2
  Interventions: Behavioral: Non-exercise activity
- B, 75% (Experimental): The investigators will compare the physical activity just-in-Time Adaptive Interventions (JITAI) to an active control working memory task within participants.There will be 4 triggers in total. Ratio intervention / active control = 3:1
  Interventions: Behavioral: Non-exercise activity
- C, 25% (Experimental): Intervention for the control group (healthy participants) is the same as for the other groups. We will compare the physical activity just-in-Time Adaptive Interventions (JITAI) to an active control working memory task within participants. There will be 4 triggers in total. Ratio intervention / active control = 1:3
  Interventions: Behavioral: Non-exercise activity

INTERVENTIONS:
Behavioral: Non-exercise activity — The 5-week intervention to assess the effects of non-exercise activity on the activity-subjective energy association incorporates two high-intensity Ambulatory Assessment (AA) weeks at the beginning and end, with a tapered 3-week Ecological Momentary Intervention (EMI) phase in between. Momentary targeted micro interventions (JITAIs) with a Within-Person-Encouragement Design (WPED) are used to tailor the activity to the individual situation and phenotype of each participant.

SUMMARY:
This approach utilizes accelerometry to measure NEA and electronic diaries for real-time psychological assessments, overcoming limitations of traditional methods such as retrospective bias and low ecological validity. Brief episodes of physical activity in daily life, which are distinctly different from structured exercise sessions, are generally linked to improved affective well-being. Notably, feelings of energy are particularly associated with incidental, unstructured, and non-exercise activities. Clinically, psychomotor retardation and diminished mood are key diagnostic features of MDD, with evidence suggesting that lower motor activity differentiates MDD patients from controls and that increased activity correlates with treatment response. In this context, the MASE project aims to design personalized BA interventions that focus on increasing NEA and, in turn, enhancing subjective energy levels to reduce depressive symptoms and prevent relapse.

DETAILED DESCRIPTION:
Mental health problems are increasing worldwide. Major depressive disorder (MDD) is considered the worldwide leading source of disability. Therapeutic approaches are not fully understood and still improvable.

Behavioral activation (BA), a successful therapeutic approach for nearly 50 years, increases activation by means of establishing short, and rewarding experiences in patients' daily life, e.g., taking a shower. Current research clearly supports the effects of BA on MDD when comparing it to no intervention. However, BA alone is not superior to other specific forms of psychotherapy. To improve BA, it is necessary to better understand the behavioral and neurobiological underpinnings. Most recently, researchers identified a new potential starting point for treating MDD: the momentary relationship between physical activity and feelings of energy in everyday life. While past research focused on exercise for treating MDD, newer studies have found that not sports (e.g., jogging) but everyday physical activity (e.g., walking stairs) improves energy. The investigators call this relationship ASEA (real-life physical activity-subjective energy association), which describes how people feel more energized and awake when moving. Secondly, we determined a specific region in the brain for ASEA and its relationship to mental health. ASEA is important from a clinical perspective: Reductions in physical activity and loss of energy symptoms affect patients most and even individuals with a history of MDD show reduced physical activity. Short interventions in patients' daily life tackling ASEA are likely to improve MDD prevention and treatment. However, it is unclear who (e.g., patients with specific brain properties) benefits most from which intervention (type of nonexercise activity, timing, location, context). For example, people with a certain brain structure may especially profit from a short slow walk with others in the morning to increase energy and reduce depression while people with another certain brain area may benefit from fast stair-climbing in the evening. Therefore, the investigators aim to a) apply brain network analyses to identify types of brains likely to profit from ASEA, (b) use artificial intelligence to identify where and when nonexercise activity helps people with certain brain properties, (c) conduct an experimental study to test if the intervention suggestions found in step (a) and (b) really work out in everyday life and (d) develop and design a smartphone app that delivers ASEA interventions and provides suggestions when and where to engage in which short nonexercise activity to maximize participation rates. In sum, the aim is to advance scientifically proven interventions by unraveling the neurobiological aspects and to tailor interventions to individuals for prevention and treatment of MDD.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient knowledge of the German language
* Written informed consent.
* Score > 15 on the Montgomery Asberg Depression rating scale (MADRS) for MDD group.
* Remission within the past year and exhibit a MADRS score < 10 for at least one month for rMDD group

Exclusion Criteria:

* Pregnancy at baseline
* Claustrophobia
* Pacemaker
* Artificial heart valves
* Active implants
* Other psychiatric disorders
* Acute suicidality, change of medication / psychotherapy during the intervention (not dosage but substance).
* For healthy participants: history of any mental health condition or first-degree relative with affective / psychotic disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change of real-life physical activity-subjective energy association | pre-post intervention (at 5 weeks)
  Subjective energy following target contexts will be assessed using the subscale Energetic Arousal from the MDMQ (VAS; scale from 0 to 100, with higher scores indicating higher energy levels).

SECONDARY OUTCOMES:
Change / stability in depressive symptoms in acute / remitted MDD patients | pre-post intervention (at 5 weeks)
  Depression severity will be evaluated using the MADRS on a 7-point Likert-scale (with higher scores indicating more depressive symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Reichert, Prof, Study Director — Department of Sport and Exercise Science University of Salzburg
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
To facilitate data sharing, the investigators (Is) will include a standardized data request form and contact information for data requests in the MASE OSF folder. Pseudonymized processed data will be suitable for sharing with research organizations that will comply with the research project's data protection policy, GDPR and relevant ethical principles. In accordance with these policies, the Is will create a standardized data sharing agreement to be used by research organizations who wish to use the data for research purposes. The legal and ethical grounds for data sharing of pseudonymized data is consent of the participant. Raw location data will never be shared externally and will never leave UB and RUB. When sharing data, the Is will include a detailed codebook on all variables, defining their type, scale, content, and if applicable their calculation. The codebook will also contain information on the methodology of data collection and on all data preprocessing steps.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Embargo on collected data until the manuscripts on the main aims of the project are accepted for publication.
Access Criteria: request form to PI (Prof. Markus Reichert)

REFERENCES:
- [Background] Reichert M, Braun U, Gan G, Reinhard I, Giurgiu M, Ma R, Zang Z, Hennig O, Koch ED, Wieland L, Schweiger J, Inta D, Hoell A, Akdeniz C, Zipf A, Ebner-Priemer UW, Tost H, Meyer-Lindenberg A. A neural mechanism for affective well-being: Subgenual cingulate cortex mediates real-life effects of nonexercise activity on energy. Sci Adv. 2020 Nov 6;6(45):eaaz8934. doi: 10.1126/sciadv.aaz8934. Print 2020 Nov. PMID 33158875
- [Background] Reichert M, Braun U, Lautenbach S, Zipf A, Ebner-Priemer U, Tost H, Meyer-Lindenberg A. Studying the impact of built environments on human mental health in everyday life: methodological developments, state-of-the-art and technological frontiers. Curr Opin Psychol. 2020 Apr;32:158-164. doi: 10.1016/j.copsyc.2019.08.026. Epub 2019 Sep 9. PMID 31610407
- [Background] Reichert M, Tost H, Reinhard I, Schlotz W, Zipf A, Salize HJ, Meyer-Lindenberg A, Ebner-Priemer UW. Exercise versus Nonexercise Activity: E-diaries Unravel Distinct Effects on Mood. Med Sci Sports Exerc. 2017 Apr;49(4):763-773. doi: 10.1249/MSS.0000000000001149. PMID 27824691
- [Background] Schmiedek F, Neubauer AB. Experiments in the Wild: Introducing the Within-Person Encouragement Design. Multivariate Behav Res. 2020 Mar-Apr;55(2):256-276. doi: 10.1080/00273171.2019.1627660. Epub 2019 Jul 2. PMID 31264902
- [Background] Abdoli N, Salari N, Darvishi N, Jafarpour S, Solaymani M, Mohammadi M, Shohaimi S. The global prevalence of major depressive disorder (MDD) among the elderly: A systematic review and meta-analysis. Neurosci Biobehav Rev. 2022 Jan;132:1067-1073. doi: 10.1016/j.neubiorev.2021.10.041. Epub 2021 Nov 4. PMID 34742925
- [Background] Biagianti B, Foti G, Di Liberto A, Bressi C, Brambilla P. CBT-informed psychological interventions for adult patients with anxiety and depression symptoms: A narrative review of digital treatment options. J Affect Disord. 2023 Mar 15;325:682-694. doi: 10.1016/j.jad.2023.01.057. Epub 2023 Jan 20. PMID 36690081
- [Background] Furukawa TA, Suganuma A, Ostinelli EG, Andersson G, Beevers CG, Shumake J, Berger T, Boele FW, Buntrock C, Carlbring P, Choi I, Christensen H, Mackinnon A, Dahne J, Huibers MJH, Ebert DD, Farrer L, Forand NR, Strunk DR, Ezawa ID, Forsell E, Kaldo V, Geraedts A, Gilbody S, Littlewood E, Brabyn S, Hadjistavropoulos HD, Schneider LH, Johansson R, Kenter R, Kivi M, Bjorkelund C, Kleiboer A, Riper H, Klein JP, Schroder J, Meyer B, Moritz S, Bucker L, Lintvedt O, Johansson P, Lundgren J, Milgrom J, Gemmill AW, Mohr DC, Montero-Marin J, Garcia-Campayo J, Nobis S, Zarski AC, O'Moore K, Williams AD, Newby JM, Perini S, Phillips R, Schneider J, Pots W, Pugh NE, Richards D, Rosso IM, Rauch SL, Sheeber LB, Smith J, Spek V, Pop VJ, Unlu B, van Bastelaar KMP, van Luenen S, Garnefski N, Kraaij V, Vernmark K, Warmerdam L, van Straten A, Zagorscak P, Knaevelsrud C, Heinrich M, Miguel C, Cipriani A, Efthimiou O, Karyotaki E, Cuijpers P. Dismantling, optimising, and personalising internet cognitive behavioural therapy for depression: a systematic review and component network meta-analysis using individual participant data. Lancet Psychiatry. 2021 Jun;8(6):500-511. doi: 10.1016/S2215-0366(21)00077-8. Epub 2021 May 3. PMID 33957075
- [Background] Heinz A, Kiefer F, Smolka MN, Endrass T, Beste C, Beck A, Liu S, Genauck A, Romund L, Banaschewski T, Bermpohl F, Deserno L, Dolan RJ, Durstewitz D, Ebner-Priemer U, Flor H, Hansson AC, Heim C, Hermann D, Kiebel S, Kirsch P, Kirschbaum C, Koppe G, Marxen M, Meyer-Lindenberg A, Nagel WE, Noori HR, Pilhatsch M, Priller J, Rietschel M, Romanczuk-Seiferth N, Schlagenhauf F, Sommer WH, Stallkamp J, Strohle A, Stock AK, Winterer G, Winter C, Walter H, Witt S, Vollstadt-Klein S, Rapp MA, Tost H, Spanagel R. Addiction Research Consortium: Losing and regaining control over drug intake (ReCoDe)-From trajectories to mechanisms and interventions. Addict Biol. 2020 Mar;25(2):e12866. doi: 10.1111/adb.12866. Epub 2019 Dec 20. PMID 31859437
- [Background] Kanning MK, Ebner-Priemer UW, Schlicht WM. How to Investigate Within-Subject Associations between Physical Activity and Momentary Affective States in Everyday Life: A Position Statement Based on a Literature Overview. Front Psychol. 2013 Apr 29;4:187. doi: 10.3389/fpsyg.2013.00187. eCollection 2013. PMID 23641221
- [Background] Liu S, Haucke M, Gross R, Schneider K, Shin J, Arntz F, Bach P, Banaschewski T, Beste C, Deserno L, Ebner-Priemer U, Endrass T, Ganz M, Ghadami A, Giurgiu M, Heinz A, Kiefer F, Kliegl R, Lenz B, Marciniak MA, Meyer-Lindenberg A, Neubauer AB, Rapp M, Smolka MN, Strehle J, Spanagel R, Spitta G, Tost H, Walter H, Zech H, Reichert D, Reichert M. Real-time mechanism-based interventions for daily alcohol challenges: Protocol for ecological momentary assessment and intervention. Digit Health. 2025 Jan 22;11:20552076241311731. doi: 10.1177/20552076241311731. eCollection 2025 Jan-Dec. PMID 39845518
- [Background] Simmonds-Buckley M, Kellett S, Waller G. Acceptability and Efficacy of Group Behavioral Activation for Depression Among Adults: A Meta-Analysis. Behav Ther. 2019 Sep;50(5):864-885. doi: 10.1016/j.beth.2019.01.003. Epub 2019 Jan 29. PMID 31422844
- [Background] Timm I, Giurgiu M, Ebner-Priemer U, Reichert M. The Within-Subject Association of Physical Behavior and Affective Well-Being in Everyday Life: A Systematic Literature Review. Sports Med. 2024 Jun;54(6):1667-1705. doi: 10.1007/s40279-024-02016-1. Epub 2024 May 6. PMID 38705972
- [Background] Tindall L, Mikocka-Walus A, McMillan D, Wright B, Hewitt C, Gascoyne S. Is behavioural activation effective in the treatment of depression in young people? A systematic review and meta-analysis. Psychol Psychother. 2017 Dec;90(4):770-796. doi: 10.1111/papt.12121. Epub 2017 Mar 16. PMID 28299896
- [Background] Torous J, Lipschitz J, Ng M, Firth J. Dropout rates in clinical trials of smartphone apps for depressive symptoms: A systematic review and meta-analysis. J Affect Disord. 2020 Feb 15;263:413-419. doi: 10.1016/j.jad.2019.11.167. Epub 2019 Dec 3. PMID 31969272
- [Background] Trull TJ, Ebner-Priemer U. Ambulatory assessment. Annu Rev Clin Psychol. 2013;9:151-76. doi: 10.1146/annurev-clinpsy-050212-185510. Epub 2012 Nov 13. PMID 23157450